CLINICAL TRIAL: NCT03261492
Title: Partnering for PA in Early Childhood: Sustainability Via Active Garden Education
Brief Title: Sustainability Via Active Garden Education
Acronym: SAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 5U01MD010667 (NIH)
Record Dates: First submitted 2017-04-13; First posted 2017-08-25 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The investigators will identify, recruit, and randomize ECEC to the SAGE intervention or a child safety attention comparison. After 16 weeks, intervention and comparison will cross over, allowing us to continue to investigate longitudinal and carry over effects. One ECEC of each pair will be randomized to the SAGE intervention and the other to the child safety attention comparison. ECEC will cross over and receive the treatment that they did not receive to ensure that all ECEC receive both curriculums.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (Experimental): SAGE curriculum is a garden-based PA and nutrition educational program and presently includes 12 lessons that can be delivered once or twice a week. The SAGE garden-based curriculum includes active games and discussion as well as activities that include watering the ECEC garden.
  Interventions: Behavioral: Physical Activity
- Child Safety Attention Comparison (Active Comparator): The goal of this comparison group is to provide centers with an engaging, useful, carefully sequenced, and easy-to-deliver curriculum so that randomization to this group does not influence attrition or reach and serves as a placebo (unlikely to affect outcomes of interest. The curriculum will include concepts and lessons for educating young children on fire, pedestrian, water, household, neighborhood and playground safety. The curriculum includes handouts, coloring sheets, comic books, games, and songs that can be implemented with minimal training and preparation.
  Interventions: Behavioral: Child Safety Attention Comparison

INTERVENTIONS:
Behavioral: Physical Activity — SAGE curriculum is a garden-based PA and nutrition educational program for early care and education centers.
  Other Names: SAGE Garden Based Curriculum
  Arms: Physical Activity
Behavioral: Child Safety Attention Comparison — The goal of this comparison group is to provide centers with an engaging, useful, carefully sequenced, and easy-to-deliver curriculum so that randomization to this group does not influence attrition or reach and serves as a placebo (unlikely to affect outcomes of interest).
  Arms: Child Safety Attention Comparison

SUMMARY:
The goal of SAGE is to determine if a garden-based curriculum can increase physical activity and improve nutrition in young children at early care and education centers (ECEC) throughout Phoenix

DETAILED DESCRIPTION:
SAGE will be delivered over a four month period using a cluster randomized controlled trial adapted crossover design, along with testing a sustainability action plan (SAP) at the organizational level. In this study, the investigators will determine the efficacy of the SAGE intervention on health in 3-4 year-old children. This study will pair match and randomize 20 ECEC from neighborhoods with high proportions of Hispanic or Latino residents. ECEC will receive either the SAGE intervention or the safety attention comparison. Then, ECEC will cross over and receive the treatment that they did not receive to ensure that all ECEC receive both curricula. The investigators will determine improvement in accelerometry measured PA and sedentary behaviors, fruit and vegetable consumption and explore eating in the absence of hunger compared to those in a child safety attention comparison. The investigators will explore secondary impacts on parenting practices that promote PA and fruit and vegetable consumption, home fruit and vegetable availability and improved household food security. This study will explore the process of delivery of the SAGE intervention on dimensions of reach, adoption, and implementation. This study will also develop, implement, and evaluate a SAP in the SAGE arm to determine replicability and institutionalization (sustainability) of the SAGE intervention and explore the relationship between of sustainability to child outcomes at follow-up. The development and success of the community Partnership and SAGE Community Advisory Board will also be evaluated using indicators of participation, representativeness, and collaboration. This study will rely on CBPR strategies and an established theoretical model to implement an engaging and translational multilevel intervention linking policy and practice. This work will test strategies for implementing IOM guidelines at the ECE level and will guide future efforts aimed at scaling up efficacious interventions for broad dissemination in vulnerable populations to reduce health disparities.

ELIGIBILITY:
ECEC Inclusion Criteria:

* Census tracts with >30% Hispanic-Latino population
* ECEC must be licensed and enroll at least 35 children aged 3-4 years old
* Space for garden install

Exclusion Criteria:

* Not participating in CACFP
* No space for a garden
* Less than 35 children aged 3-5 years old enrolled

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change physical activity; sedentary time | Four assessment periods: baseline, 4 months, 8 months weeks, and 12 months
  Assessed by ActiGraph accelerometers
fruit and vegetable consumption | Four assessment periods: baseline, 4 months, 8 months weeks, and 12 months
  24 hr diet recalls

SECONDARY OUTCOMES:
Impact on parenting practices in physical activity (PA) | Four assessment periods: baseline, 4 months, 8 months weeks, and 12 months
  Assessed by physical activity
Impact on improved home fruit and vegetable availability | Four assessment periods: baseline, 4 months, 8 months weeks, and 12 months
  Assessed by completing Home Food Inventory questionnaire
Impact on parenting practices in fruits and vegetables | Four assessment periods: baseline, 4 months, 8 months weeks, and 12 months
  Assessed by fruit and vegetable pactices questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Lee, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Mello GT, Szeszulski J, O'Connor T, Lorenzo E, Hill JL, Lee RE. Effects of Sustainability via Active Garden Education on preschool-aged children's locomotor skills. Transl Behav Med. 2025 Jan 16;15(1):ibaf052. doi: 10.1093/tbm/ibaf052. PMID 41047236
- [Derived] Szeszulski J, Lorenzo E, Todd M, O'Connor TM, Hill J, Shaibi GQ, Vega-Lopez S, Buman MP, Hooker SP, Lee RE. Early Care and Education Center Environmental Factors Associated with Product- and Process-Based Locomotor Outcomes in Preschool-Age Children. Int J Environ Res Public Health. 2022 Feb 15;19(4):2208. doi: 10.3390/ijerph19042208. PMID 35206392
- [Derived] Szeszulski J, Lorenzo E, O'Connor T, Hill JL, Shaibi GQ, Buman MP, Vega-Lopez S, Hooker SP, Lee RE. Exploring Correlates of Preschool-Aged Children's Locomotor Skills: Individual and Parent Demographics and Home Environment. Percept Mot Skills. 2021 Apr;128(2):649-671. doi: 10.1177/0031512520980938. Epub 2020 Dec 20. PMID 33342342